CLINICAL TRIAL: NCT05645887
Title: Human Albumin Treatment in Adult Septic Shock. A Study Evaluating Immune Response and Organ Failure.
Acronym: ALBUMIM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal reorganisations and lack of funding by the sponsor
Sponsor: Albimmune SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-001949-20
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Serum Albumin, Human; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Albumim (20%, 300mL, 60gr) in 180 min IV (Experimental): Further doses of albumin (60g/l) will be administered daily from day 0 to day 7 in patients with serum albumin concentrations <35 g/L.
  Interventions: Drug: Human albumin
- Saline solution 0,9% (500mL) in 180 min IV (Placebo Comparator): Saline solution will be given from day 0 to day 7.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Human albumin — Human albumin from day 0 to 7 if serum albumin concentrations <35g/l.
  Arms: Human Albumim (20%, 300mL, 60gr) in 180 min IV
Other: Saline solution — Saline solution from day 0 to day 7.
  Arms: Saline solution 0,9% (500mL) in 180 min IV

SUMMARY:
The goal of this phase 2, multicenter, randomized, controlled study is to evaluate the effect of albumin treatment on B cell and other immune cell gene exptression in adults with septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years and <85 years of age.
2. Community-acquired pneumonia, urinary, skin or biliary infection.
3. Treatment with antibiotics at least one course in the first 6 hours of suspected infection.
4. Meets Septic Shock criteria defined by the presence of sepsis with persistent hypotension despite initial adequate volume resuscitation requiring vasopressors for more than 4h to maintain MAP>65 mmHg and having a serum lactate level > 2mmol/L (18mg/L).
5. SOFA score ≥ 5 points.
6. Albumin plasma level <35g/L.
7. Lymphocytes count < 1,100 cel/mL.
8. Admitted to ICU or IMU

Exclusion Criteria:

1. Septic shock lasting for more than 24h.
2. ECMO or hemoadsortion therapy.
3. Contraindications to receive albumin.
4. Nosocomial or healthcare-associated infections (surgical intervention or hospitalization within 30 days prior to diagnosis of sepsis).
5. Chronic Renal Failure (KIDGO stage 3-5) or dialysis.
6. Liver cirrhosis.
7. A known malignancy that is progressing or has required active treatment within the past 3 months.
8. Patient with end-stage disease (unrelated to sepsis) defined as patients who prior to the current hospitalization are expected to live < 6 months (as assessed by the study physician).
9. Known New York Heart Association (NYHA) class II to IV heart failure or unstable angina, acute coronary disease or myocardial infarction within 6 months prior to diagnosis of sepsis.
10. Known immunocompromised state, including human immunodeficiency virus infection, or medication known to be immunosuppressive.
11. Participation in an interventional investigational study within 30 days prior to diagnosis of sepsis.
12. Likely to be non-compliant or uncooperative during the study (e.g. substance abuse, uncontrolled psychiatric disorder or any chronic condition that may interfere with the study).
13. Albumin administration within the last 14 days.
14. Subjects with severe neurological or severe head trauma disorders.
15. Pregnant and/or breast-feeding woman.
16. Patients who cannot provide prior informed consent and when there is documented evidence that the patient has no legal surrogate decision marker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
1.1 Evaluate B cell response to albumin treatment | at day 0
  Measured by the Immunology Complex (Discovery Study).
1.2 Evaluate B cell response to albumin treatment | at day 1
  Measured by the Immunology Complex (Discovery Study).
1.3 Evaluate B cell response to albumin treatment | at day 3
  Measured by the Immunology Complex (Discovery Study).
1.4 Evaluate B cell response to albumin treatment | at day 7
  Measured by the Immunology Complex (Discovery Study).
1.5 Evaluate B cell response to albumin treatment | at day 14
  Measured by the Immunology Complex (Discovery Study).
1.6 Evaluate other immune cell response to albumin treatment | at day 0
  Measured by the Immunology Complex (Discovery Study).
1.7 Evaluate other immune cell response to albumin treatment | at day 1
  Measured by the Immunology Complex (Discovery Study).
1.8 Evaluate other immune cell response to albumin treatment | at day 3
  Measured by the Immunology Complex (Discovery Study).
1.9 Evaluate other immune cell response to albumin treatment | at day 7
  Measured by the Immunology Complex (Discovery Study).
1.10 Evaluate other immune cell response to albumin treatment | at day 14
  Measured by the Immunology Complex (Discovery Study).

SECONDARY OUTCOMES:
1.1. Identify additional biomarkers of the immune response to albumin treatment. | at day 0, 1, 3, 7 and 14.
  Measured by the IGCGS score.
1.2.1 Evaluate the functionality of antibody-secreting B cells. | at day 0, 1, 3, 7 and 14.
  Measurated by B cell function.
1.2.2 Evaluate the functionality of antibody-secreting B cells. | at day 0, 1, 3, 7 and 14.
  Measurated by serum immunoglobilin levels (g/L).
1.2.3 Evaluate the functionality of antibody-secreting B cells. | at day 0, 1, 3, 7 and 14.
  Measurated by glycosylation.
1.2.4 Evaluate the functionality of antibody-secreting B cells. | at day 0, 1, 3, 7 and 14.
  Measurated by blood immunophenotyping.
2.1To further investigate the mechanisms of albumin treatment on the immune system. | at day 0, 1, 3, 7 and 14.
  Measurated by assessment of whole blood RNA sequencing.
2.2 To further investigate the mechanisms of albumin treatment on the immune system. | at day 0, 1, 3, 7 and 14.
  Measurated by assessment of single-cell RNA sequencing.
2.3 To further investigate the mechanisms of albumin treatment on the immune system. | at day 0, 1, 3, 7 and 14.
  Measurated by assessment of CITE-seq.
2.4 To further investigate the mechanisms of albumin treatment on the immune system. | at day 0, 1, 3, 7 and 14.
  Measurated by assessment of immunophenotyping of B cells by high-dimensional spectral flow cytometry.
3. Evaluate whether albumin activates B cells at the mucosal interface. | at day 0, 3, 7 and 14.
  Measurated by assessment of circulating levels of immunoglobulins and glycosylated immunoglobulins.
4.1. Evaluate the effect of albumin treatment on systemic inflammation. | at day 0, 1, 3, 7 and 14.
  Measurated by plasma cytokines: IL-1β, IL-1ra, IL-6, IL-7, IL-8, IL-10, IL-17, TNF-α, TNFr1, IFN-γ, MCP-1, MCP-3, RAGE.
4.2.1 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by sCr (mg/dL).
4.2.2 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by urine output.
4.2.3 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by balance fluid.
4.2.4 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by KDIGO stage 2-3.
4.2.5 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by TIMP-2.
4.2.6 Evaluate kidney. | at day 0, 1, 3, 7 and 14.
  Measurated by IGFBP 7.
4.3.1 To explore the effect of albumin on gut mucosa immunoglobulins. | at day 0, 3, 7 and 14.
  Measurated by composition of bacterial communities bound to IgA.
4.3.2 To explore the effect of albumin on gut mucosa immunoglobulins. | at day 0, 3, 7 and 14.
  Measurated by composition of whole fecal bacteria.
4.3.3 To explore the effect of albumin on gut mucosa immunoglobulins. | at day 0, 3, 7 and 14.
  Measurated by antibody-binding profile of microbes.
4.3.4 To explore the effect of albumin on gut mucosa immunoglobulins. | at day 0, 3, 7 and 14.
  Measurated by bacterial reactivity of peripheral blood antibodies.
5.1 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by angiopoeitin 1.
5.2 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by angiopoeitin 2.
5.3 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by MR-proADM.
5.4 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by Selectin.
5.5 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by VCAM-1.
5.6 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by ICAM-1.
5.7 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by endothelin-1.
5.8 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by thrombomodulin.
5.9 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by syndecan 1-4.
5.10 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by prot C (mg/L).
5.11 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by heparan sulfate.
5.12 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by VEGF.
5.13 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by sphingosine-1-phosphate (S1P).
5.14 Evaluate the effect of albumin on endothelial and glycocalix function. | at day 0, 1, 3, 7 and 14.
  Measurated by PAI-1.
6.1 Time on vasopressors. | 14 days
  Measurated by time on vasopressors.
6.2 Time on mechanical ventilation. | 14 days
  Measurated by time on mechanical ventilation.
6.3 Time on renal replacement. | 14 days
  Measurated by time on renal replacement.
7. Proportion of patients with secondary infections. | 90 days
  Measurated by the number of patients with secondary infections.
8.1. Proportion of patients dead at 28 and 90 days. | 90 days
  Measurated by the number of patients dead at 28 and 90 days.
8.2. Proportion of patients re-admitted to ICU at 28 days. | 28 days
  Measurated by the number of re-admitted to UCI at 28 days.
8.3. Proportion of re-hospitalized patients at 28 days. | 28 days
  Measurated by the number of re-hospitalized patients at 28 days.
8.4.1 Evaluate the sequential SOFA score. | at day 0, 1, 3, 7 and 14.
  Measurated by SOFA score.
8.4.2 Evaluate the sequential APACHE II score. | at day 0, 1, 3, 7 and 14.
  Measurated by APACHE II score.
8.4.3 Evaluate the sequential TISS-28 score. | at day 0, 1, 3, 7 and 14.
  Measurated by TISS-28 score.
9. Evaluate quality of life (QoL) at day 90. | At day 0 and 90
  Measurated by the EQ-5D-5L questionnaire.
10. Proportion of participants with any AEs related to albumin treatment, SAEs and SUSARs. | 90 days
  Measured by the number of AE, SAEs and SUSARS presented by the participants.